CLINICAL TRIAL: NCT05334511
Title: Effects Of Functional Electrical Stimulation On Functional Rehabilitation In Children With Erb's Palsy
Brief Title: Functional Electrical Stimulation On Functional Rehabilitation In Children With Erb's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/RCR &AHS/21/0701
Record Dates: First submitted 2022-04-02; First posted 2022-04-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Erb's Palsy
MeSH Terms: conditions — Brachial Plexus Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Electrical Stimulation (Experimental): functional electrical stimulation with Frequency 20 pps with Pulse width of 300 msec.
  Interventions: Other: Functional Electrical Stimulation

INTERVENTIONS:
Other: Functional Electrical Stimulation — functional electrical stimulation with Frequency 20 pps with Pulse width of 300 msec.

SUMMARY:
Erb's palsy is a type of brachial plexus injury occurs in infants due to injury of nerves during childbirth. Injury causes weakness or paralysis of different muscles. Different type of approaches are made for the treatment of erb;s palsy such passive range of motion, stretching ,splinting ,electrotherapy etc. In erb's palsy the most affected ranges are shoulder abduction and shoulder external rotation. Quasi experimental study will be done on the patient with erb's palsy intervention applied will be functional electrical stimulation (a low frequency current) applied 5 day a weeks for 2 weeks than on alternate days for the rest of the treatment. Setting for functional electrical stimulation will be Frequency 20 pps with Pulse width of 300 msec. 18 patient will be recruited . "Assumed population standard deviation"4.24" "Confidence level""0.95" "Acceptable error""2". Pre-intervention reading will be taken on modified mallet scale and universal goniometer and post intervention measurement will be taken after 02, 04 ,06 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Erb's Palsy
* Children of age 15 months to 3 years

Exclusion Criteria:

* hemiplegic cerebral palsy
* children with upper limb fractures
* obstetrical brachial plexus injury
* upper limb contracture

Ages: 15 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Modified mallet scale Score | Baseline, 2nd, 4th and 6th Months
  Modified Mallet scale evaluation of function and arm appearance. In addition to assessing the classical shoulder functions of the classical Modified Mallet system, supination and the resting position are evaluated. In the resting position, medial rotation at the shoulder is scored on a scale of 1 to 5. 1 is the lowest score and 5 is the highest score
Change in range of motion | Baseline, 2nd, 4th and 6th months
  A goniometer is an instrument that measures the available range of motion at a joint. The art and science of measuring the joint ranges in each plane of the joint are called goniometry.
  To measure the range of motion physical therapists most commonly use a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Children Complex Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okafor UA, Akinbo SR, Sokunbi OG, Okanlawon AO, Noronha CC. Comparison of electrical stimulation and conventional physiotherapy in functional rehabilitation in Erb's palsy. Nig Q J Hosp Med. 2008 Oct-Dec;18(4):202-5. doi: 10.4314/nqjhm.v18i4.45029. PMID 19391320
- [Background] Nath RK, Somasundaram C. Significant improvement in nerve conduction, arm length, and upper extremity function after intraoperative electrical stimulation, neurolysis, and biceps tendon lengthening in obstetric brachial plexus patients. J Orthop Surg Res. 2015 Apr 19;10:51. doi: 10.1186/s13018-015-0191-y. PMID 25895832
- [Background] Huang X, Jiang Z, Sun H, Xie B, Lu F, Huang W, Wang T, Xiong H. The effect of a high-quality nursing model employing low-frequency pulse electrical stimulation combined with early systemic functional exercises on the function of the affected limb in brachial plexus injury patients. Am J Transl Res. 2021 May 15;13(5):4939-4948. eCollection 2021. PMID 34150078
- [Background] Elnaggar RK. Shoulder Function and Bone Mineralization in Children with Obstetric Brachial Plexus Injury After Neuromuscular Electrical Stimulation During Weight-Bearing Exercises. Am J Phys Med Rehabil. 2016 Apr;95(4):239-47. doi: 10.1097/PHM.0000000000000449. PMID 26829088